CLINICAL TRIAL: NCT00157014
Title: Clinical and Laboratory Evaluation of Acute Rejection, Myocyte Growth, Repair, and Oxidative Stress Following de Novo Cardiac Transplant: A Comparison Between Tacrolimus- and Cyclosporine- Based Immunoprophylactic Regimens With MPA TDM
Brief Title: Canadian Cardiology de Novo Study: A Comparison Between Tacrolimus- and Cyclosporine- Based Immunoprophylactic Regimens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKC-009
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Heart Diseases; Heart Transplantation
Keywords: Antirejection; Treatment Outcome; Immunosuppression; Treatment Effectiveness; Anti-rejection therapy
MeSH Terms: conditions — Heart Diseases | interventions — Tacrolimus; Cyclosporine; Mycophenolic Acid; Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tacrolimus - Adult (Experimental): Adults: 0.05 - 0.10 mg/ kg/ day in 2 divided doses starting within 10 days of transplant
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Methylprednisolone; Drug: Prednisone
- Cyclosporine - Adult (Active Comparator): Adults: 3-5 mg/ kg/ day in 2 divided doses starting within 10 days of transplant
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Methylprednisolone; Drug: Prednisone
- Tacrolimus - Pediatric (Experimental): Pediatrics: 0.05 - 0.30 mg/ kg/ day in 2-3 divided doses starting within 10 days of transplant
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Methylprednisolone; Drug: Prednisone
- Cyclosporine - Pediatric (Active Comparator): Pediatrics: 6 - 10 mg/ kg/ day in 2-3 divided doses starting within 10 days of transplant
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus — Oral
  Other Names: Prograf; FK506
  Arms: Tacrolimus - Adult; Tacrolimus - Pediatric
Drug: Cyclosporine — Oral
  Arms: Cyclosporine - Adult; Cyclosporine - Pediatric
Drug: Mycophenolate mofetil — Intravenous and Oral
  Other Names: CellCept
Drug: Methylprednisolone — Intravenous
Drug: Prednisone — Oral

SUMMARY:
The purpose of this study is to assess the safety and efficacy of tacrolimus in de novo heart transplantation.

DETAILED DESCRIPTION:
Subcellular markers will be assessed in relationship to cellular acute rejection in de novo cardiac transplant recipients receiving either tacrolimus or cyclosporine as their primary immunosuppressant

Two parallel active arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or their legal guardians) who are capable of understanding, and who have been fully informed of the purpose of the study and the risks of participation.
* Patients (or their legal guardians) who have signed and dated the Informed Consent form and are willing and able to follow the study protocol.
* Patients who are primary cadaveric heart transplant recipients.
* Males or females from birth.
* Female patients of child-bearing potential who have a current negative pregnancy test and agree to practice effective birth control, as judged by the investigator, while participating in the study. Prepubescent pediatric patients will not require pregnancy testing.
* Patients able to tolerate oral medication and who do not have a gastrointestinal condition likely to affect the absorption kinetics or metabolism of the oral study medications.

Exclusion Criteria:

* Previous organ transplant recipients.
* Multi-organ transplant recipients.
* Recipients of a heart from a donor with incompatible ABO blood type.
* Patients with significant graft dysfunction and/or significant de novo infection(s) at time of randomization
* Patients with known hypersensitivity to tacrolimus, cyclosporine, mycophenolate mofetil (MMF), daclizumab, prednisone, cremophor, polysorbate 80 and/or polyoxyl 60 hydrogenated castor oil (HCO-60).
* Patients who are pregnant or lactating or planning to become pregnant prior to completion of the study.
* Patients who have consumed an investigational product in the 30 days prior to transplantation or at any time during post-transplantation follow-up.
* Patients receiving cholestyramine or colestipol.
* Patients having any one of the following at enrolment:

  1. History of malignancy, not chart-documented as cured or active malignancy (with exception of eradicable non-metastatic in-situ basal cell or squamous cell carcinoma).
  2. Leukopenia (white cell count < 2500/cu mm).
  3. Anemia (hemoglobin < 80 g/L).
  4. Positive test for hepatitis B surface antigen and/or hepatitis C.
  5. Historical positive test for human immunodeficiency virus (HIV).
  6. Serum creatinine > 230 umol/l.
  7. Continual elevation of AST and/or ALT to >= 3X the upper limit of normal.
  8. Body mass index (weight in kg/height in m2) > 30.
* Undiagnosed diabetes mellitus as determined by 2 hour (2h) oral glucose tolerance test (OGTT) or fasting glucose test or uncontrolled diabetes mellitus at screening. In either case, the patient may be declared as no longer excluded by this criterion upon establishment of control of the diabetes through appropriate medical management.
* Blood glucose >= 11.1 mmol/L at pre-operative assessment.
* Patients having a significant disease, substance dependency, or disability that may prevent adherence to, or understanding of, the protocol and/or the investigator's instructions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2004-05-10 (Actual); Primary Completion 2008-07-18 (Actual); Study Completion 2008-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Canada, Inc.
Locations (10):
- Los Angeles, California, United States
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec

REFERENCES:
- See also: Link to Prescribing Information — http://www.astellas.us/docs/prograf.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * 3 patients randomized to cyclosporine actually received tacrolimus and were included in the Treatment Exposure Population for tacrolimus.
  * 2 patients randomized for tacrolimus were excluded from Treatment Exposure Population - 1 never received drug; 1 received incorrect drug without a waiver.
Period: Overall Study
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Started | 52 | 46 | 5 | 6
Completed | 45 | 41 | 4 | 5
Not Completed | 7 | 5 | 1 | 1
Not completed — Death | 4 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Medications withdrawn on family request | 0 | 1 | 0 | 0
Not completed — Patient withdrawn by investigator | 1 | 0 | 0 | 0
Not completed — Patient unable to return in nursing home | 1 | 0 | 0 | 0
Not completed — Patient would not receive transplant | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult | Tacrolimus - Pediatric | Cyclosporine - Pediatric | Total
Number analyzed (Participants) | 52 | 46 | 5 | 6 | 109
Age, Customized [Number; unit: Participants]
  0 - ˂ 2 Years | 0 | 0 | 1 | 1 | 2
  2 - 10 Years | 0 | 0 | 1 | 2 | 3
  10 - ˂ 18 Years | 0 | 0 | 3 | 3 | 6
  18 - 49 Years | 14 | 18 | 0 | 0 | 32
  50 - 59 Years | 18 | 15 | 0 | 0 | 33
  60 - 69 Years | 18 | 12 | 0 | 0 | 30
  70 Years and Older | 2 | 1 | 0 | 0 | 3
Sex/Gender, Customized [Number; unit: Participants]
  Male | 43 | 37 | 0 | 2 | 82
  Female | 9 | 9 | 5 | 4 | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  European descent/ White | 48 | 40 | 5 | 4 | 97
  Black | 2 | 4 | 0 | 1 | 7
  East Indian | 2 | 0 | 0 | 1 | 3
  Latin American | 0 | 1 | 0 | 0 | 1
  Aboriginal | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Markers of Growth, Apoptosis, Inflammation and Oxidation Measured in Endomyocardial Biopsies
Description: The markers assessed were p-ERK ½ (phosphorylated extracellular signal-regulated kinase), p-JNK (phosphorylated jun N-terminal kinase) and p-p38 MAPK (phosphorylated mitogen-activated protein kinase).
  The data for each biopsy marker were expressed as a ratio of its densitometry / densitometry of glyceraldehyde-3-phosphate dehydrogenase (GAPDH).
  Change is defined as Week 52 assessment- Week 2 assessment.
Time Frame: 2 Weeks and 52 Weeks
Population: The number of participants analyzed per arm represents Treatment Exposure Population- defined as all patients receiving at least 1 dose of study medication summarized according to treatment received regardless of randomization allocation.
Measure: Mean (Standard Deviation); unit: Densitometry / Densitometry of GAPDH
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Densitometry / Densitometry of GAPDH
  p-ERK ½ - Week 2: number analyzed (Participants) | 36 | 37
  p-ERK ½ - Week 2 | 0.70 (0.500) | 0.90 (0.641)
  p-ERK ½ - Week 52: number analyzed (Participants) | 30 | 27
  p-ERK ½ - Week 52 | 0.87 (0.539) | 0.79 (0.674)
  p-ERK ½ - Change from Week 2: number analyzed (Participants) | 26 | 25
  p-ERK ½ - Change from Week 2 | 0.05 (0.834) | -0.05 (0.662)
  p-JNK - Week 2: number analyzed (Participants) | 36 | 37
  p-JNK - Week 2 | 1.10 (0.813) | 1.23 (0.722)
  p-JNK - Week 52: number analyzed (Participants) | 30 | 27
  p-JNK - Week 52 | 1.33 (0.890) | 1.46 (0.792)
  p-JNK - Change from Week 2: number analyzed (Participants) | 26 | 25
  p-JNK - Change from Week 2 | 0.03 (1.188) | 0.22 (0.957)
  p-p38 MAPK - Week 2: number analyzed (Participants) | 35 | 37
  p-p38 MAPK - Week 2 | 0.48 (0.450) | 0.54 (0.556)
  p-p38 MAPK - Week 52: number analyzed (Participants) | 28 | 27
  p-p38 MAPK - Week 52 | 0.63 (0.664) | 0.77 (0.717)
  p-p38 MAPK - Change from Week 2: number analyzed (Participants) | 25 | 25
  p-p38 MAPK - Change from Week 2 | 0.14 (0.733) | 0.23 (0.828)

2. Primary Outcome: The Change in the Markers of Growth, Apoptosis, Inflammation and Oxidation Measured in Endomyocardial Biopsies (Pediatric Population)
Description: The markers assessed were p-ERK ½, p-JNK and p-p38 MAPK.
  The data for each biopsy marker were expressed as a ratio of its densitometry / densitometry of glyceraldehyde-3-phosphate dehydrogenase (GAPDH).
  Change is defined as Week 52 assessment- Week 2 assessment.
Time Frame: 2 Weeks and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Densitometry / Densitometry of GAPDH
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
Densitometry / Densitometry of GAPDH
  p-ERK ½ - Week 2: number analyzed (Participants) | 3 | 5
  p-ERK ½ - Week 2 | 1.74 (0.972) | 1.67 (0.682)
  p-ERK ½ - Week 52: number analyzed (Participants) | 2 | 4
  p-ERK ½ - Week 52 | 0.93 (0.184) | 1.22 (0.633)
  p-ERK ½ - Change from Week 2: number analyzed (Participants) | 1 | 3
  p-ERK ½ - Change from Week 2 | -0.09 (0) | -0.27 (0.309)
  p-JNK - Week 2: number analyzed (Participants) | 3 | 5
  p-JNK - Week 2 | 1.17 (0.420) | 0.91 (0.430)
  p-JNK - Week 52: number analyzed (Participants) | 2 | 4
  p-JNK - Week 52 | 0.57 (0.085) | 0.82 (0.537)
  p-JNK - Change from Week 2: number analyzed (Participants) | 1 | 3
  p-JNK - Change from Week 2 | -0.21 (0) | 0.04 (0.189)
  p-p38 MAPK - Week 2: number analyzed (Participants) | 3 | 5
  p-p38 MAPK - Week 2 | 0.83 (0.467) | 0.43 (0.364)
  p-p38 MAPK - Week 52: number analyzed (Participants) | 2 | 4
  p-p38 MAPK - Week 52 | 0.24 (0.014) | 0.58 (0.432)
  p-p38 MAPK - Change from Week 2: number analyzed (Participants) | 1 | 3
  p-p38 MAPK - Change from Week 2 | -0.04 (0) | 0.34 (0.630)

3. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: MCP-1
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  MCP-1= monocyte chemoattractant protein-1
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
pg/mL
  Pre-Transplant: number analyzed (Participants) | 48 | 44
  Pre-Transplant | 233.05 (292.832) | 193.63 (144.696)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 229.96 (263.084) | 180.90 (145.067)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | 42.92 (165.517) | -16.49 (126.586)

4. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: s-ICAM
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  s-ICAM= soluble-intracellular adhesion molecule
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
ng/mL
  Pre-Transplant: number analyzed (Participants) | 50 | 45
  Pre-Transplant | 766.58 (449.572) | 674.46 (429.036)
  Week 52: number analyzed (Participants) | 41 | 40
  Week 52 | 590.30 (369.942) | 503.71 (305.531)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 41 | 40
  Change from Pre-Transplant at Week 52 | -227.58 (366.136) | -183.96 (250.382)

5. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: E-selectin
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
ng/mL
  Pre-Transplant: number analyzed (Participants) | 50 | 43
  Pre-Transplant | 90.40 (72.801) | 98.96 (89.153)
  Week 52: number analyzed (Participants) | 41 | 40
  Week 52 | 68.60 (51.911) | 80.93 (70.383)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 41 | 40
  Change from Pre-Transplant at Week 52 | -18.58 (48.247) | -19.16 (52.080)

6. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: Homocysteine
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
μmol/L
  Pre-Transplant: number analyzed (Participants) | 50 | 44
  Pre-Transplant | 14.2 (6.94) | 15.9 (6.97)
  Week 52: number analyzed (Participants) | 40 | 40
  Week 52 | 13.5 (4.19) | 15.8 (5.33)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 40 | 40
  Change from Pre-Transplant at Week 52 | 0.3 (5.02) | 0.7 (7.61)

7. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: hsCRP
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  hsCRP= high-sensitivity C Reactive Protein
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
mg/L
  Pre-Transplant: number analyzed (Participants) | 49 | 45
  Pre-Transplant | 32.85 (50.859) | 21.83 (33.547)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 3.01 (3.313) | 3.95 (5.273)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | -34.32 (54.257) | -18.69 (35.354)

8. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: F2 Isoprostanes
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
pg/mL
  Pre-Transplant: number analyzed (Participants) | 48 | 45
  Pre-Transplant | 52.03 (76.090) | 53.94 (78.476)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 30.08 (25.905) | 50.44 (68.416)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | -13.29 (40.543) | -3.43 (103.457)

9. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: T-bars
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  T-bars = thiobarbituric acid reactive substances
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
nmol/mL
  Pre-Transplant: number analyzed (Participants) | 50 | 45
  Pre-Transplant | 3.78 (1.586) | 3.91 (2.059)
  Week 52: number analyzed (Participants) | 40 | 39
  Week 52 | 3.25 (1.365) | 3.14 (1.198)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 40 | 39
  Change from Pre-Transplant at Week 52 | -0.64 (1.724) | -0.77 (2.182)

10. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: Nitrotyrosine
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
nM
  Pre-Transplant: number analyzed (Participants) | 50 | 45
  Pre-Transplant | 422.63 (393.554) | 482.43 (390.702)
  Week 52: number analyzed (Participants) | 41 | 39
  Week 52 | 451.88 (443.372) | 368.95 (262.693)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 41 | 39
  Change from Pre-Transplant at Week 52 | 71.44 (332.351) | -99.79 (228.268)

11. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: GSH/GSSG
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  GSH/GSSG= ratio of reduced to oxidised glutathione
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Ratio
  Pre-Transplant: number analyzed (Participants) | 49 | 45
  Pre-Transplant | 55.07 (62.780) | 58.83 (71.289)
  Week 52: number analyzed (Participants) | 39 | 38
  Week 52 | 51.69 (55.721) | 53.72 (55.264)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 39 | 38
  Change from Pre-Transplant at Week 52 | -2.07 (70.036) | -5.55 (80.490)

12. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: BNP
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  BNP= Brain Natriuretic Peptide
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
ng/L
  Pre-Transplant: number analyzed (Participants) | 49 | 44
  Pre-Transplant | 4314.8 (4861.78) | 4240.8 (4673.72)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 670.1 (1053.21) | 1856.8 (5077.26)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | -4018.4 (5043.28) | -1446.7 (6460.33)

13. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: Troponin T
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
ug/L
  Pre-Transplant: number analyzed (Participants) | 49 | 44
  Pre-Transplant | 0.30 (0.686) | 0.28 (0.878)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 0.03 (0.116) | 0.04 (0.120)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | -0.32 (0.768) | -0.27 (0.958)

14. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: Osteopontin
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
ng/mL
  Pre-Transplant: number analyzed (Participants) | 50 | 44
  Pre-Transplant | 11.88 (9.528) | 11.14 (12.278)
  Week 52: number analyzed (Participants) | 41 | 38
  Week 52 | 8.77 (10.462) | 10.49 (8.987)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 41 | 38
  Change from Pre-Transplant at Week 52 | -2.22 (10.615) | 0.20 (11.158)

15. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: Fibrinogen
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
g/L
  Pre-Transplant: number analyzed (Participants) | 48 | 44
  Pre-Transplant | 4.4 (1.27) | 4.4 (1.23)
  Week 52: number analyzed (Participants) | 40 | 40
  Week 52 | 3.4 (0.87) | 3.8 (0.77)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 40 | 40
  Change from Pre-Transplant at Week 52 | -1.1 (1.48) | -0.5 (1.23)

16. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: IL-6
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
  IL= Interleukin
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
pg/mL
  Pre-Transplant: number analyzed (Participants) | 48 | 45
  Pre-Transplant | 3.36 (4.221) | 2.54 (3.159)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 0.98 (0.743) | 0.90 (0.651)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | -2.84 (4.635) | -1.56 (3.146)

17. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: IL-18
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
pg/mL
  Pre-Transplant: number analyzed (Participants) | 48 | 45
  Pre-Transplant | 574.0 (291.89) | 496.2 (246.90)
  Week 52: number analyzed (Participants) | 40 | 40
  Week 52 | 534.6 (290.38) | 427.2 (217.07)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 40 | 40
  Change from Pre-Transplant at Week 52 | 5.2 (289.66) | -71.0 (243.81)

18. Secondary Outcome: Changes in Circulating Markers of Inflammation, Oxidation, Growth, Apoptosis, Differentiation and Survival: Cystatin-C
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment.
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
mg/L
  Pre-Transplant: number analyzed (Participants) | 49 | 45
  Pre-Transplant | 1.21 (0.414) | 1.29 (0.490)
  Week 52: number analyzed (Participants) | 42 | 40
  Week 52 | 1.29 (0.533) | 1.48 (0.714)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 42 | 40
  Change from Pre-Transplant at Week 52 | 0.06 (0.464) | 0.27 (0.744)

19. Secondary Outcome: Number of Acute Rejection Episodes by International Society of Heart and Lung Transplantation (ISHLT) Criteria
Description: Acute rejection was defined as a rejection with ISHLT Grade ≥3A or by the presence of hemodynamic compromise.
  ISHLT Grades ≥3A include: Multifocal Moderate Rejection; Diffuse, Borderline Severe Acute Rejection; and Severe Acute Rejection.
  Patients may report more than one acute rejection.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: Rejection Episodes
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Rejection Episodes
  Total Acute Rejection Episodes | 8 | 8
  Acute Rejection Episodes with ISHLT Grade ≥3A | 3 | 7
  Acute Rejection Episodes w/ Hemodynamic Compromise | 6 | 2

20. Secondary Outcome: Time to First Acute Rejection Episode Following de Novo Cardiac Transplant
Description: Acute Rejection was defined as a rejection with ISHLT Grade ≥3A or by the presence of hemodynamic compromise.
  ISHLT Grades ≥3A include: Multifocal Moderate Rejection; Diffuse, Borderline Severe Acute Rejection; and Severe Acute Rejection.
  Time to first acute rejection is defined as: date of onset - date of transplant.
Time Frame: 52 Weeks
Population: The population analyzed represents Treatment Exposure Population- defined as all patients receiving at least 1 dose of study medication summarized according to treatment received regardless of randomization allocation. Only participants who experienced acute rejection were included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 6 | 8
Days | 55.0 (35.60) | 35.60 (132.86)

21. Secondary Outcome: Number of Patients Requiring Antilymphocyte Antibodies or Steroids for Treatment of Severe Acute Rejection
Description: Severe Acute Rejection is defined as rejection with ISHLT Grade 4.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Patients | 0 | 0

22. Secondary Outcome: Number of Cardiac Rejection Episodes Requiring Treatment
Description: The number of rejection episodes requiring treatment (medications started/ stopped, non-medication treatment, or both) regardless of biopsy grade or presence of hemodynamic compromise.
Time Frame: 52 Weeks
Population: The number of participants analyzed per arm represents Treatment Exposure Population - defined as all patients receiving at least 1 dose of study medication summarized according to treatment received regardless of randomization allocation.
Measure: Number; unit: Rejection Episodes
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Rejection Episodes | 12 | 11

23. Secondary Outcome: Mean Cases of Acute Rejection (MCAR) Per Patient
Description: MCAR represents the average number of acute rejections among all patients in each treatment group. Results were based on rejection episodes with endomyocardial biopsies.
  Acute rejection was defined as a rejection with ISHLT Grade ≥3A or by the presence of hemodynamic compromise.
  ISHLT Grades ≥3A include: Multifocal Moderate Rejection; Diffuse, Borderline Severe Acute Rejection; and Severe Acute Rejection.
Time Frame: 52 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: MCAR per patient
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
MCAR per patient | 0.15 (0.46) | 0.17 (0.38)
Statistical Analysis 1: Comparison: Tacrolimus - Adult vs Cyclosporine - Adult; Test type: Superiority or Other; p = 0.4725, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons were performed

24. Secondary Outcome: Number of Patients With Successful Steroid Taper or Withdrawal at Weeks 26 and 52
Description: A successful steroid taper or withdrawal was defined as steroids (prednisone) being discontinued or tapered to the suggested dose level after week 26.
Time Frame: 26 Weeks and 52 Weeks
Population: as for outcome 22
Measure: Number; unit: Patients
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Patients
  Week 26 | 22 | 16
  Week 52 | 33 | 29

25. Secondary Outcome: Number of Patients With Treatment Failure and Crossover for Treatment Failure
Description: Treatment failure was defined as death, re-transplantation, withdrawal due to an Adverse Event, or a switch of main immunosuppressant medication, whichever came first.
  Crossover was defined as a switch from originally administered primary immunosuppressant (tacrolimus or cyclosporine) to the alternate primary immunosuppressant.
Time Frame: 52 Weeks
Population: as for outcome 22
Measure: Number; unit: Patients
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult
Number analyzed (Participants) | 52 | 46
Patients
  Treatment Failures | 6 | 11
  Crossover for Treatment Failures | 2 | 8

26. Secondary Outcome: Changes in Circulating Markers of Inflammation and Oxidation: F2 Isoprostanes (Pediatric Population)
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
pg/mL
  Pre-Transplant: number analyzed (Participants) | 5 | 5
  Pre-Transplant | 106.06 (37.974) | 104.68 (53.812)
  Week 52: number analyzed (Participants) | 3 | 4
  Week 52 | 69.71 (38.620) | 66.48 (33.298)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 3 | 4
  Change from Pre-Transplant at Week 52 | -38.31 (47.563) | -30.07 (80.246)

27. Secondary Outcome: Changes in Circulating Markers of Inflammation and Oxidation: Nitrotyrosine (Pediatric Population)
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
nM
  Pre-Transplant: number analyzed (Participants) | 5 | 5
  Pre-Transplant | 233.08 (211.491) | 12701.21 (21666.231)
  Week 52: number analyzed (Participants) | 3 | 4
  Week 52 | 5462.99 (7988.134) | 41147.62 (37565.740)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 3 | 4
  Change from Pre-Transplant at Week 52 | 5148.42 (7849.554) | 21514.62 (49626.968)

28. Secondary Outcome: Changes in Circulating Markers of Inflammation and Oxidation: hsCRP (Pediatric Population)
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
mg/L
  Pre-Transplant: number analyzed (Participants) | 5 | 4
  Pre-Transplant | 30.46 (32.274) | 12.08 (14.771)
  Week 52: number analyzed (Participants) | 3 | 4
  Week 52 | 26.31 (45.109) | 2.43 (1.348)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 3 | 4
  Change from Pre-Transplant at Week 52 | -7.85 (78.126) | -13.94 (16.461)

29. Secondary Outcome: Changes in Circulating Markers of Inflammation and Oxidation: Cystatin-C (Pediatric Population)
Description: Change is defined as Week 52 assessment - Pre-Transplant assessment
Time Frame: Pre-Transplant and 52 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
mg/L
  Pre-Transplant: number analyzed (Participants) | 5 | 4
  Pre-Transplant | 0.86 (0.248) | 0.77 (0.194)
  Week 52: number analyzed (Participants) | 3 | 4
  Week 52 | 0.87 (0.133) | 0.84 (0.111)
  Change from Pre-Transplant at Week 52: number analyzed (Participants) | 3 | 4
  Change from Pre-Transplant at Week 52 | -0.11 (0.197) | -0.01 (0.108)

30. Secondary Outcome: Number of Acute Rejection Episodes by International Society of Heart and Lung Transplantation (ISHLT) Criteria (Pediatric Population)
Description: Acute rejection was defined as a rejection with ISHLT Grade ≥3A or by the presence of hemodynamic compromise.
  ISHLT Grades ≥3A include: Multifocal Moderate Rejection; Diffuse, Borderline Severe Acute Rejection; and Severe Acute Rejection.
  Patients may report more than one rejection episode.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: Rejection Episodes
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
Rejection Episodes
  Total Acute Rejection Episodes | 3 | 3
  Acute Rejection Episodes with ISHLT Grade ≥3A | 3 | 3
  Acute Rejection Episodes w/ Hemodynamic Compromise | 0 | 0

31. Secondary Outcome: Time to First Acute Rejection Episode Following de Novo Cardiac Transplant (Pediatric Population)
Description: as for outcome 20
Time Frame: 52 Weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 3 | 3
Days | 56.3 (27.06) | 49.0 (15.62)

32. Secondary Outcome: Number of Patients Requiring Antilymphocyte Antibodies or Steroids for Treatment of Severe Acute Rejection (Pediatric Population)
Description: Severe Acute Rejection was defined as rejection with ISHLT Grade 4.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
Patients | 0 | 0

33. Secondary Outcome: Number of Cardiac Rejection Episodes Requiring Treatment (Pediatric Population)
Description: A summary of rejection episodes requiring treatment regardless of biopsy grade or presence of hemodynamic compromise.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: Rejection Episodes
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
Rejection Episodes | 3 | 3

34. Secondary Outcome: Mean Cases of Acute Rejection (MCAR) Per Patient (Pediatric Population)
Description: as for outcome 23
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: MCAR per patient
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
MCAR per patient | 0.60 (0.55) | 0.50 (0.55)
Statistical Analysis 1: Comparison: Tacrolimus - Pediatric vs Cyclosporine - Pediatric; Test type: Superiority or Other; p = 0.8373, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons were performed

35. Secondary Outcome: Number of Patients With Successful Steroid Taper or Withdrawal at Weeks 26 and 52 (Pediatric Population)
Description: as for outcome 24
Time Frame: 26 Weeks and 52 Weeks
Population: as for outcome 22
Measure: Number; unit: Patients
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
Patients
  Week 26 | 2 | 3
  Week 52 | 1 | 1

36. Secondary Outcome: Number of Patients With Treatment Failure and Crossover for Treatment Failure (Pediatric Population)
Description: as for outcome 25
Time Frame: 52 Weeks
Population: as for outcome 22
Measure: Number; unit: Patients
Arm/Group | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Number analyzed (Participants) | 5 | 6
Patients
  Treatment Failures | 1 | 3
  Crossover for Treatment Failures | 0 | 3

ADVERSE EVENTS:
Time Frame: After the initiation of study drug up to 30 days after the last dose of study drug.
Description: Treatment Emergent Adverse Events were reported.
  Within a preferred term, patients were counted once.
Arm/Group | Tacrolimus - Adult | Cyclosporine - Adult | Tacrolimus - Pediatric | Cyclosporine - Pediatric
Serious Adverse Events (participants affected / at risk) | 21/52 | 24/46 | 3/5 | 5/6
Other Adverse Events (participants affected / at risk) | 52/52 | 46/46 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus - Adult (N=52) | Cyclosporine - Adult (N=46) | Tacrolimus - Pediatric (N=5) | Cyclosporine - Pediatric (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 2 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 2 | 1 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Adrenal mass (Endocrine disorders) | 0 | 1 | 0 | 0
Blindness cortical (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter related complication (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Heart transplant rejection (Immune system disorders) | 2 | 1 | 0 | 0
Transplant rejection (Immune system disorders) | 2 | 1 | 0 | 0
American trypanosomiasis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1
Haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 3 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0
Inferior vena caval occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 1 | 0 | 0
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus - Adult (N=52) | Cyclosporine - Adult (N=46) | Tacrolimus - Pediatric (N=5) | Cyclosporine - Pediatric (N=6)
Aneamia (Blood and lymphatic system disorders) | 18 | 15 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 9 | 9 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 12 | 9 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 4 | 0 | 0
Atrial flutter (Cardiac disorders) | 3 | 3 | 0 | 0
Bradycardia (Cardiac disorders) | 6 | 3 | 0 | 0
Fluid overload (Cardiac disorders) | 4 | 6 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 2 | 0 | 0
Oedema due to cardiac disease (Cardiac disorders) | 3 | 4 | 0 | 0
Oedema peripheral (Cardiac disorders) | 6 | 14 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 6 | 0 | 0
Pericardial effusion (Cardiac disorders) | 5 | 6 | 1 | 0
Pulmonary oedema (Cardiac disorders) | 3 | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 4 | 3 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 3 | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Becker's muscular dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Amblyopia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 13 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 26 | 8 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 15 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 9 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 5 | 2 | 0 | 0
Chest pain (General disorders) | 4 | 2 | 0 | 0
Chills (General disorders) | 1 | 3 | 0 | 0
Fatigue (General disorders) | 2 | 7 | 0 | 0
Hyperthermia (General disorders) | 2 | 4 | 0 | 0
Influenza like illness (General disorders) | 3 | 0 | 0 | 0
Oedema peripheral (General disorders) | 14 | 6 | 0 | 2
Pyrexia (General disorders) | 4 | 4 | 0 | 2
Oedema (General disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 4 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 3 | 0 | 0
Influenza (Infections and infestations) | 1 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 6 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 0 | 0
Staphylococcal infection (Infections and infestations) | 4 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 1 | 2
Urinary tract infection (Infections and infestations) | 6 | 2 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper repiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 5 | 3 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 5 | 0 | 0
Cardiac murmur (Investigations) | 3 | 3 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 4 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 1 | 0
Weight increased (Investigations) | 10 | 9 | 1 | 0
Cytomegalovirus antigen positive (Investigations) | 0 | 0 | 0 | 1
Epstein-Barr virus antibody positive (Investigations) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 11 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 4 | 2 | 0
Gout (Metabolism and nutrition disorders) | 2 | 5 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 7 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 8 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 4 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 4 | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 6 | 4 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 8 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 3 | 0 | 0
Headache (Nervous system disorders) | 11 | 13 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 3 | 0 | 0
Tremor (Nervous system disorders) | 23 | 13 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 4 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 5 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 1 | 0 | 0
Depression (Psychiatric disorders) | 6 | 5 | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 12 | 0 | 1
Renal failure (Renal and urinary disorders) | 11 | 12 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 4 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 3 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 3 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 6 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 7 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Removal of foreign body (Surgical and medical procedures) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 21 | 26 | 3 | 4
Hypotension (Vascular disorders) | 13 | 7 | 0 | 0

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.